CLINICAL TRIAL: NCT06919861
Title: A Randomized, Double-blind, Two-group Crossover Study Comparing the Pharmacokinetics, Pharmacodynamics, and Safety of Nanokine (Nanogen) With Eprex® (Janssen-Cilag Ltd) in Healthy Male Volunteers
Brief Title: Pharmacokinetics, Pharmacodynamics, and Safety of Nanokine Produced by Nanogen Pharmaceutical Joint Stock Company
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanogen Pharmaceutical Biotechnology Joint Stock Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NNG31
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Natural Blood and Blood Product Toxicity
MeSH Terms: interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanokine 4000 IU (Experimental): Nanokine 4000 IU, prefilled syringe, subcutaneous injection. Nanokine 4000 IU will be transported and handed over to the Study Center by the Sponsor. Nanokine 4000 IU should be stored in a refrigerator of 2-8°C.
  Interventions: Biological: Erythropoietin alfa
- Eprex 4000 IU (Active Comparator): Eprex 4000 IU, pre-closed syringe, subcutaneous injection. Eprex 4000 IU will be transported and handed over directly to the Study Center by the supplier (with a contract with the Sponsor).
  Eprex 4000 IU should be stored in a refrigerator of 2- 8 °C.
  Interventions: Biological: Erythropoietin alfa

INTERVENTIONS:
Biological: Erythropoietin alfa — Experimental drug: Nanokine 4000 IU, prefilled syringe, subcutaneous injection Manufactured: Nanogen Biopharmaceutical JSC.
  Arm 1 (22 volunteers): Nanokineinjection 4000 IU will be administered subcutaneously on Day 1, and after a 28-day washout period, Eprex® injection 4000 IU will be administered subcutaneously on Day 29.
  Other Names: Nanokine
Biological: Erythropoietin alfa — Comparator drug: Eprex® 4000 IU, prefilled syringe, subcutaneous injection Manufactured: Janssen-Cilag Ltd
  Arm 2 (22 volunteers): Eprex® injection 4000 IU will be administered subcutaneously on Day 1, and after a 28-day washout period, Eprex injection 4000 IU will be administered subcutaneously on Day 29.
  Total: 44 participants will be recruited in the trial.
  Other Names: Eprex

SUMMARY:
This clinical trial aims to compare the pharmacokinetic (PK), pharmacodynamic (PD) parameters, and safety between Nanokine of Nanogen Pharmaceutical Joint Stock Company and Eprex® of Janssen Cilag Ltd on healthy male volunteers.

The biosimilarity of erythropoietin (EPO) between Nanokine (test) and Eprex® (comparator) was evaluated in a randomized, double-blind, two-sequence, crossover study.

Subjects received a 4,000 IU subcutaneous dose of either formulation, followed by the alternate after a 28-day washout.

Key pharmacokinetic (PK) parameters, Cmax and AUCinf, were assessed, with geometric mean ratios/GMR (90% CI) falling within the regulatory range (0.80-1.25). Pharmacodynamic (PD) markers (reticulocyte count, hematocrit, hemoglobin, and RBC count) need to show comparable effects.

Safety evaluation (adverse events and serious adverse events, other safety assessments such as vital signs, testing, and examination) supports their interchangeability in clinical use.

DETAILED DESCRIPTION:
Erythropoietin (EPO) is a glycoprotein hormone essential for red blood cell (RBC) formation, primarily produced in the kidneys. Recombinant human erythropoietin (rHuEPO) or erythropoiesis-stimulating agents (ESAs) are used to treat anemia in chronic renal failure, chemotherapy-induced anemia, and to reduce transfusion needs in surgery.

Nanokine, currently considered as a follow-on biological product of Eprex® developed by Nanogen Biopharmaceutical JSC, is produced in CHO cells. This study evaluates the bioequivalence of Nanokine and Eprex® in healthy volunteers, comparing pharmacokinetics (PK), pharmacodynamics (PD), and safety.

A randomized, double-blind, single-dose, two-sequence crossover trial was conducted in 44 healthy male volunteers (19-45 years, BMI 18.0-27.0 kg/m²). Participants received a 4,000 IU subcutaneous injection of either Eprex® or Nanokine, followed by the alternate after a 28-day washout. Blood samples for PK analysis were taken at multiple time points up to 144 hours postdose, while PD markers (reticulocyte count, hematocrit, hemoglobin, RBC count) were measured up to 312 hours postdose.

This study is conducted at the Center for Clinical Pharmacology-Hanoi Medical University, following the Vietnam guideline of Biomedical research, ethical, and regulatory guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Male aged between 18 and 45.
* Weight between 50 kg and 70 kg, BMI between 18 and 27 at the time of screening.
* Subjects of reproductive age must approve the use of effective contraception (such as oral contraceptives, intrauterine or implantable, intrauterine placement, physical methods, etc.) from screening until 6 months after the last dose.
* Signed an informed consent form to participate in the study.

Exclusion Criteria:

Subjects who meet at least one of the following criteria will be excluded from the study:

* Use EPO (erythropoietin), darbepoetin, or another source of EPO protein, immunoglobulin, within 3 months before screening.
* History of severe allergic reactions or anaphylactic reactions to biological products.
* There are any clinically significant diseases such as high blood pressure, other cardiovascular diseases, psychiatry, cancer, acute and chronic respiration, diabetes, chronic inflammation (such as rheumatoid arthritis, lupus erythematosus, etc.), or autoimmune diseases.
* Having a history of red blood cell diseases such as thalassemia, sickle cell...
* Those who bled over 400mL or donated blood within 8 weeks of the scheduled first dose.
* People with screening results:

  * Hemoglobin level below 12 g/dL or above 17 g/dL;
  * Vitamin B12 level below 200 pg/mL;
  * Ferritin level below 21.8 ng/mL;
  * Transferrin level below 190 mg/dL;
  * Albumin level below 3.5 g/dL or more than 4.8 g/dL;
  * Reticulocyte, erythrocytes, platelets, or serum potassium level over the normal range
  * Positive on the HIV antibody, HBsAg, HCV(Hepatitis C Virus) antibody tests.
  * Those whose vital signs are measured in the sitting position after resting for over 3 minutes meet more than one of the following: Systolic BP below 90mmHg or over 160mmHg, Diastolic BP below 50mmHg or over 100mmHg, Pulse rate over 100.
* History of drug abuse, or tested positive in the urine drug screening
* Those who have a drinking problem or are unable to abstain from alcohol during the study period.
* Those who have smoked over 10 cigarettes daily on average for the last 3 months or who can't renounce smoking during the trial period.
* People who have ingested caffeine-containing food within 3 days of the scheduled first dose or who can't abstain from the during the trial period.
* Those with peculiar eating habits or who can't have meals provided by the study center.
* Those who participated in other clinical trials and were administered other study drugs within 1 year of the scheduled first dose.
* Those who are preparing for pregnancy or who do not agree with contraception during the trial period

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
AUC0-inf | 10 minutes before administration (day 1/day 29); 1, 2, 4, 6, 8, 10, 12, 14,16, 24, 36, 48, 72, 96, 120, 144 hrs after administration for each period]
  Area under the plasma concentration versus time curve from time 0 to infinity
Cmax | 10 minutes before administration (day 1/day 29); 1, 2, 4, 6, 8, 10, 12, 14,16, 24, 36, 48, 72, 96, 120, 144 hrs after administration for each period]
  Peak plasma concentration

SECONDARY OUTCOMES:
AUClast | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  Area Under Curve last
Clast.obs | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  Concentration above the last observed quantitative threshold
Tmax | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  Time of maximum concentration of Erythropoietin
T1/2 | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  Terminal half-life(t1/2) of Erythropoietin: Time (hours) required for the serum drug concentration to be reduced by half
Tlast | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  The last time at which the observed concentration is above the quantitative threshold.
CL.obs | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  Apparent clearance
Vz.obs | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  Apparent volume of distribution
Lambda.z | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  The rate of elimination corresponds to the final half-life
TEmax | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  Time to maximum reticulocyte count (TEmax).
ΔEmax | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  Maximum increase in observed reticulocyte count compared to pre-dose
ΔAUEC0-inf | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  Area under the effect curve of increased reticulocyte count from time 0 to infinity
Hemoglobin | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  Hemoglobin (Hb)
Hematocrit | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  Hematocrit (Hct)
RBC count | 10 minutes before administration (day 1/day 29); 12, 24, 48, 72, 96, 120, 144, 216, 312 hrs after administration for each period]
  Red blood cells count
Adverse events | Baseline to 312 hours after the crossover dose
  Adverse events (AE); Serious adverse events (SAE); Other safety assessments such as vital signs, testing, and examination.